CLINICAL TRIAL: NCT00243763
Title: Phase 1 Dose Escalating Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of TKI258 in Subjects With Refractory or Relapsed Multiple Myeloma
Brief Title: TKI258 in Subjects With Refractory or Relapsed Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTKI258A2103
Record Dates: First submitted 2005-10-21; First posted 2005-10-25 (Estimated); Last update posted 2009-11-23 (Estimated); Status verified 2009-11

CONDITIONS: Multiple Myeloma
Keywords: Refractory Multiple Myeloma or; Relapsed Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one

INTERVENTIONS:
Drug: TKI258

SUMMARY:
The primary objective of this study is to determine the maximum tolerated dose (MTD), dose limiting toxicity (DLT), and safety profile of CHIR-258 when administered to subjects with refractory or relapsed multiple myeloma (MM).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of multiple myeloma
* Evidence of relapsed or refractory disease

Exclusion Criteria:

* Intracranial disease or epidural disease
* Clinically significant cardiac disease
* Diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose
Dose limiting toxicity
Safety profile

SECONDARY OUTCOMES:
Evaluation of pharmacokinetics and pharmacodynamics

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis
Locations (5):
- United States (5):
  - Mayo Clinic - Arizona, Scottsdale, Arizona
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic - Minnesota, Rochester, Minnesota

REFERENCES:
- [Derived] Wang X, Kay A, Anak O, Angevin E, Escudier B, Zhou W, Feng Y, Dugan M, Schran H. Population pharmacokinetic/pharmacodynamic modeling to assist dosing schedule selection for dovitinib. J Clin Pharmacol. 2013 Jan;53(1):14-20. doi: 10.1177/0091270011433330. Epub 2013 Jan 24. PMID 23400739